CLINICAL TRIAL: NCT01325896
Title: Maintenance Treatment of Multiple Myeloma (MM) After Autologous Peripheral Blood Transplant (PBSCT) Using Polyethylene Glycol alpha2B Interpheron (PEG-INTRON)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Collaborators: Haematology Service, (Unknown)
Responsible Party: Dr Adrián Alegre Amor., Hematology Service, Hospital Universitario de La Princesa. Madrid, Spain
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI-MM-01
Record Dates: First submitted 2011-03-11; First posted 2011-03-30 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Multiple Mieloma
Keywords: Multiple Mieloma, PEG-Intron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients are receiving PEG-Intron (Other)
  Interventions: Drug: PEG-Intron sc injection

INTERVENTIONS:
Drug: PEG-Intron sc injection — This program is only open to patients with multiple myeloma who have achieved a complete or partial response after a myelosuppressive chemotherapy regimen followed by autologous stem cell infusion of peripheral blood transplant (PBSCT) as treatment intensification. These patients will be treated with PEG-Intron as maintenance therapy, to be permitted during the same concomitant administration of corticosteroids and / or bisphosphonates.
  PEG-Intron: 35 mcg per week by subcutaneous injection to progression or recurrence of the disease, or for 5 years maximum.
  Patients were administered PEG-Intron to a uniform dose of 15 mg initial week for 2 weeks. If this dose is tolerated, it would be gradually increased to 25 mg and then to 35 mg every 2 weeks, assuming that there is no toxicity of grade 3 or worse.

SUMMARY:
* Multiple myeloma accounts for approximately 1% of all cancers and 10% of hematologic malignancies. Between 50 and 70% of symptomatic patients presented response to induction chemotherapy. The rate of complete responses (CR) achieved with standard induction of these treatments is less than 5% of cases and the median event-free survival between 2 and 3 years although most of the patients died from the disease.
* High dose chemotherapy with autologous stem cell transplant has improved the response rate and survival of patient with MM. However eventually all patients relapse with a median EFS between 40-50 months post-transplant.
* To improve these results and sustain remission, various maintenance treatment have been proposed as is the case of Interpheron alpha2b s.c. (Intron A) that has shown benefits in a meta-analysis.
* Intron A s.c. need administration of 3 days per week and is not well tolerated
* Recently a new formulation of Interpheron alpha2b is available. Conjugated with polietilenglicol (Pegintron) that need only one dose weekly and has not been tested in MM.
* The purpose of this study is to evaluate the role of Pegintron as maintenance after autologous transplant in MM

ELIGIBILITY:
Inclusion Criteria:

* Patients ≤ 65 years old diagnosed with multiple myeloma in stage II or III of Durie-Salmon staging.
* Patients who have achieved a complete response, partial after a myelosuppressive chemotherapy treatment followed by infusion of peripheral blood progenitor cells as first-line treatment. The criteria used to define the complete or partial response are the EBMT, ABMTR IBMTR and set out in the criteria paper of Bladé J, Samson D, Reece D, et al 1998
* Subjects must have a Karnofsky performance status ≥ 60% at the time of joining the program.
* Subjects must have adequate renal and hepatic function, defined as <2 times the upper limit of normal laboratory.
* Subjects must have adequate hematologic function, defined as: platelets> 50,000/μl, ≥Hemoglobin 9.0 g/dl, total leukocyte account> 2.000/μl
* No history of any cancer within the past 5 years except squamous cell carcinoma or basal cell skin or cervical carcinoma in stage I or in situ.
* No history of hypersensitivity to interferon alfa or any other part of the injection.
* No severe clotting disorders, thrombophlebitis or pulmonary embolism, or decompensated liver disease.
* Pregnant or lactating at the time of diagnosis can not participate in this therapeutic program. During the same, men and women participants should not conceive children. Also, women who become pregnant will be withdrawn from the protocol.
* Obtaining informed consent.

Exclusion Criteria:

* Patients > 65 years old.
* Patients with multiple myeloma stage I of Durie-Salmon staging system.
* Patients who have not achieved a complete or partial response after a myelosuppressive chemotherapy regimen followed by infusion of progenitor cells from peripheral blood autologous treatment of any kind is allowed intensification of chemotherapy and pretransplant conditioning regimen. The criteria used to define the complete or partial response are the EBMT, ABMTR IBMTR and set out in the criteria paper of Bladé J, Samson D, Reece D, et al 1998
* Treatment with any investigational drug within 30 days prior to the addition to this protocol.
* Subjects with severe cardiovascular disease.
* Subjects with a history of neuropsychiatric disorder that requires hospitalization.
* Subjects with thyroid dysfunction or uncontrolled diabetes mellitus (refractory to treatment).
* Subjects with active infection and / or uncontrolled.
* Pregnant or lactating women or women of childbearing age not practicing effective contraception.
* Patients with previous psychiatric disease, especially moderate or severe depression or a history of severe psychiatric disorder, including psychosis, suicidal thoughts or suicide attempts. In severe depression cover the following points: (a) hospitalization for depression (b) electroconvulsive therapy for depression or (c) depression leading to the prolonged absence at work or to alter significantly the daily functions. Can be consider the entrance into the study of subjects with mild depression, where it is demonstrated by pre-treatment assessment individual's emotional state is clinically stable and in which case a treatment program formulated for the patient who will become part of the patient's medical record.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2002-09; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Time to Progression (TTP) and WHO (World Health Organization) Toxicity scale | three years
  Evaluate the number of Participants with Adverse Events, and provide guidelines for treatment with PEG-Intron (either in association with corticosteroids and / or bisphosphonate), administered weekly to patients with multiple myeloma who have achieved a complete or partial response after a myelosuppressive chemotherapy regimen, followed by an infusion of autologous peripheral blood progenitor cell (PBSCT) as treatment intensification.

SECONDARY OUTCOMES:
Increase of Response (anti-tumoral effect) and Dose Tolerance | three years
  Evaluate the anti-tumor efficacy of this maintenance treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adrián Alegre Amor, Physician Doctor, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; José García Laraña, Physician, Principal Investigator — Hospital Ramón y Cajal. Madrid, Spain; Juan José Lahuerta, Physician Doctor, Principal Investigator — Hospital 12 de Octubre. Madrid, Spain; Jesús San Miguel, Physician Doctor, Principal Investigator — Hospital Clínico Universitario. Salamanca, Spain
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Madrid, Spain

REFERENCES:
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033
- [Background] Bjorkstrand B, Svensson H, Goldschmidt H, Ljungman P, Apperley J, Mandelli F, Marcus R, Boogaerts M, Alegre A, Remes K, Cornelissen JJ, Blade J, Lenhoff S, Iriondo A, Carlson K, Volin L, Littlewood T, Goldstone AH, San Miguel J, Schattenberg A, Gahrton G. Alpha-interferon maintenance treatment is associated with improved survival after high-dose treatment and autologous stem cell transplantation in patients with multiple myeloma: a retrospective registry study from the European Group for Blood and Marrow Transplantation (EBMT). Bone Marrow Transplant. 2001 Mar;27(5):511-5. doi: 10.1038/sj.bmt.1702826. PMID 11313685